CLINICAL TRIAL: NCT02393183
Title: The Effect of a New Antioxidant Combination (ASTED) on Mild Thyroid Eye Disease, a Placebo Controlled Randomized Clinical Trial
Brief Title: The Effect of a New Antioxidant Combination (ASTED) on Mild Thyroid Eye Disease (TED)
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Do not access to the drug
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106955-24580-124-03-93
Record Dates: First submitted 2015-03-07; First posted 2015-03-19 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Thyroid Eye Disease
Keywords: Antioxidant; Graves' ophthalmopathy; Thyroid eye disease; Severity score; Activity score; Quality of life
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ASTED (Experimental): Antioxidant Supplements for TED (ASTED):
  to evaluate the effect of selected antioxidant vitamins and minerals supplement (Twice daily)
  1. β- Carotene (30 mg)
  2. Vit C (100 mg)
  3. Vit E (Alpha-Tocopherol Acetate): 60-200 IU
  4. Calcium phosphate dihydrate (40 mg)
  5. Zinc oxide (4 mg, elemental)
  6. Copper gluconate (3.5 mg)
  7. Sodium selenite 23 mg= Selenium 100 µg
  8. Nicotinamide (a form of vit.B3) (10 mg)
  Interventions: Drug: ASTED
- Selenium (Active Comparator): Selenium (100mic) Twice daily
  Interventions: Dietary Supplement: Selenium
- Placebo (Placebo Comparator): Placebo Twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ASTED — A tablet of ASTED will be taken twice a day
  Other Names: Antioxidant Supplement for Thyroid Eye Disease
  Arms: ASTED
Dietary Supplement: Selenium — A tablet of 100 microgram of Selenium (same shape and color) will be taken twice a day
  Arms: Selenium
Other: Placebo — A tablet of Placebo (same shape and color) will be taken twice a day
  Arms: Placebo

SUMMARY:
This randomized clinical trial is designed to evaluate the effect of selected antioxidant vitamins and minerals supplement named as ASTED:

1. β- Carotene (30 mg)
2. Vit C (100 mg)
3. Vit E (Alpha-Tocopherol Acetate): 60-200 IU
4. Calcium phosphate dihydrate (40 mg)
5. Zinc oxide (4 mg, elemental)
6. Copper gluconate (3.5 mg)
7. Sodium selenite 23 mg= Selenium 100 µg
8. Nicotinamide (a form of vit.B3) (10 mg)

in patients with mild Thyroid eye disease according to EUGOGO classification. To be given twice a day.

DETAILED DESCRIPTION:
1. To determine total eye score (NOSPECS severity score) before and after treatment in each of the three arms of the study and make a before - after as well as an inter-arm comparison.
2. To determine Score of thyroid eye disease Quality of life questionnaire (TED-QOL) before and after treatment in each of the three arms of the study and make a before - after as well as an inter-arm comparison.
3. To determine clinical activity score (CAS Score) before and after treatment in each of the three arms of the study and make a before - after as well as an inter-arm comparison.
4. To determine Serum thyroid auto-antibodies (Anti thyroid peroxidase (TPO), Anti-thyrogluboline) and Thyroid function test (Free T4, T3, and TSH) level before and after treatment in each of the three arms of the study and make a before - after as well as an inter-arm comparison.
5. To determine the rate of side effects in each arm and make a comparison.

ELIGIBILITY:
Inclusion Criteria:

1. Mild TED of less than 18 months duration (as recorded by the patient).
2. No active state (Clinical activity score of less than 3).
3. No previous specific therapy for TED, except for local measures (artificial tear, head elevation, low salt diet).
4. Euthyroidism as a result of remission after a course of antithyroid drug (ATD) therapy, or euthyroidism for at least 2 months since commencing ATD or after thyroidectomy, or euthyroidism for at least 6 months after radioiodine therapy. Hypothyroid patients after thyroidectomy or radioiodine were replaced with levothyroxine. Euthyroidism was defined as normal serum free thyroxine, total or free triiodothyronine concentrations, and thyrotropin (TSH) levels below 4 mU/Liter Patients were kept euthyroid for the whole duration of the study.
5. Age 18-70 years.

Exclusion Criteria:

1. TED severity of more than mild TED.
2. Pregnancy
3. Drug and/or alcohol abuse
4. Severe concomitant illness
5. Inability to comply with the study protocol
6. No informed consent
7. Use of selenium- or vitamin/minerals-containing preparations in the last 3 months.
8. Developing more severe TED in the course of the trial so that requires steroid treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change of total eye score (NOSPECS severity score) | 0, 3, 6 months
  Change of eye score during the study period

SECONDARY OUTCOMES:
Change of score of thyroid eye disease Quality of life questionnaire (TED-QOL) | 0, 3, 6 months
  Change of score of thyroid eye disease Quality of life during study period

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen B Kashkouli, MD, Study Director — Iran University of Medical Sciences
Locations (1):
- Rassoul Akram Hospital, Tehran, Iran